CLINICAL TRIAL: NCT02182128
Title: A Phase I Open-label Dose-escalation Study of Continuous Twice-daily Oral Treatment With BIBF 1120 in Japanese Patients With Advanced Solid Tumours
Brief Title: A Dose-escalation Study of BIBF 1120 in Japanese Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.19
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Tumors
MeSH Terms: conditions — Neoplasms | interventions — nintedanib

ARMS (1):
- BIBF 1120 (Experimental)
  Interventions: Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBF 1120

SUMMARY:
Confirmation of BIBF 1120 administered from 150 mg twice daily (b.i.d.) to 250 mg b.i.d. as safe and tolerable treatment in Japanese patients with advanced solid tumours, overall safety, pharmacokinetic parameters, biomarkers, and efficacy of BIBF 1120.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with a confirmed diagnosis of an advanced, non resectable and/or metastatic solid tumour (except for malignant lymphoma)
2. Patients who have not responded to conventional treatment, or for whom no therapy of proven efficacy was available, or who were not amenable to established forms of treatment
3. Patients recovered from any therapy-related toxicities from previous chemo-, hormone-, immuno-, or radio-therapies (except for epilation) at least over the following periods of time:

   * four weeks after chemotherapy (at least 2 weeks after receiving antimetabolite or at least 6 weeks after nitrosourea or mitomycin C)
   * two weeks after receiving hormone therapy
   * four weeks after receiving radiation therapy (2 weeks after radiation for symptom control)
   * two weeks after receiving immunotherapy
   * four weeks after surgical procedures
4. Age 20 years or older
5. Life expectancy of at least 3 months
6. Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2
7. Patients retaining a significant physiological compensatory function and without manifest marked disorders of the hematopoietic system, heart, lung, liver, kidneys, etc., i.e., patients with sufficient baseline organ function

   * An absolute neutrophil count more than 1500/mm3
   * A platelet count more than 100000/mm3
   * A haemoglobin count more than 9.0 g/dL
   * Serum creatinine less than 1.5-fold the upper limit value of the normal range
   * Bilirubin less than 1.5-fold the upper limit value of the normal range
   * Activities of aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) less than 1.5-fold the upper limit value of normal range (if related to liver metastases less than 2.5-fold the upper limit value of the normal range)
   * Saturation pulse oxygen (SpO2) level not less than 90%
8. No participation in other clinical trials within 4 weeks before start of therapy within this trial
9. Written informed consent given that is consistent with ICH-GCP guidelines

Exclusion criteria

1. Brain tumour, and/or brain metastases requiring therapy
2. History of obvious pulmonary fibrosis or interstitial pneumonitis in chest X-ray including pneumoconiosis or radiation-induced pulmonary fibrosis expanding out of radiation field
3. Patients with difficulty in swallowing study medication
4. Gastrointestinal disorders that might interfere with the absorption of the study drug (Crohn's disease, ulcerative colitis, broad resection of the stomach)
5. Patients with diarrhoea greater than CTCAE grade 2
6. Patients within 4 weeks after major surgical procedures or patients with active ulcers or with injuries with incomplete wound healing
7. History of autoimmune disease
8. History of serious drug hypersensitivity
9. History of cardiac infarction or congested heart failure of New York Heart Association Classification (NYHA) II or greater within previous 6 months
10. Serious illness or concomitant non-oncological disease difficult to be controled by medication, such as active infectious disease, hepatic failure, renal failure, pulmonary fibrosis, interstitial pneumonitis, hemorrhagic tendency, heart disease (congested heart failure, angina, arrhythmia, etc.), uncontrolled, severe hypertension, and diabetes
11. Pregnancy or breastfeeding
12. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception until 4 weeks after the last trial visit
13. Patients positive in tests of hepatitis B (HBs) antigen, hepatitis C (HCV)antibody, or HIV antibody
14. Alcohol or drug abuse
15. Patient not suitable for participation in this clinical trial in the opinion of the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-06; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) associated with increasing doses of BIBF 1120 | Up to 36 months
Incidence and intensity of Adverse Events according to Common Toxicity Criteria (CTCAE Version 3.0) associated with increasing doses of BIBF 1120 | up to 36 months

SECONDARY OUTCOMES:
maximum tolerated dose (MTD) of BIBF 1120 | Up to 36 months
Objective tumour response according to the response evaluation criteria in solid tumours (RECIST) | Up to 36 months
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 12 hours after single dose administration (AUC0-12) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 12 hours after the first drug administration
Change from baseline in peripheral blood biomarkers | Baseline, day 2, day 8, day 30
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24hours after single dose administration (AUC0-24) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after the first drug administration
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable analyte plasma concentration after single dose administration (AUC0-tz) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after the first drug administration
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity after single dose administration (AUC0-∞) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after the first drug administration
The percentage of the AUCtz-∞ that is obtained by extrapolation (%AUCtz-∞) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after the first drug administration
Maximum measured concentration of the analyte in plasma following a single dose (Cmax) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after the first drug administration
Time from dosing to the maximum concentration of the analyte in plasma following a single dose (tmax) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after the first drug administration
Terminal half-life of the analyte in plasma after single dose administration (t1/2) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after the first drug administration
Terminal rate constant in plasma after single dose administration (λz) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after the first drug administration
Mean residence time of the analyte in the body after single dose oral administration (MRTpo) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after the first drug administration
Apparent clearance of the analyte in plasma after single dose extravascular administration (CL/F) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after the first drug administration
Apparent volume of distribution during the terminal phase λz following extravascular administration (Vz/F) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after the first drug administration
Area under the concentration-time curve of the analyte in plasma at steady state over the time interval from 0 to 24hours (AUC0-24,ss) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after drug administration
Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after drug administration
Τime from last dosing to the maximum concentration of the analyte in plasma at steady state over a uniform dosing interval τ (tmax,ss) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after drug administration
Terminal half-life of the analyte in plasma at steady state (t1/2,ss) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after drug administration
Terminal rate constant in plasma at steady state (λz,ss) | Up to 36 month
Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after drug administration
Predose concentration of the analyte in plasma at steady state immediately before administration of the next dose (Cpre,ss) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after drug administration
Average concentration of the analyte in plasma at steady state (Cavg) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after drug administration
Mean residence time of the analyte in the body at steady state after oral administration (MRTpo,ss) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after drug administration
Apparent clearance of the analyte in plasma at steady state after extravascular multiple dose administration (CL/F,ss) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after drug administration
Apparent volume of distribution during the terminal phase λz at steady state following extravascular administration (Vz/F,ss) | before and 0.5, 1, 2, 3, 4, 6, 8, 10 and 24 hours after drug administration
Accumulation ratio (RA) | Up to 36 month
Predose concentration of the analyte in plasma immediately before administration of the n-th dose (Cpre,n) | Day 8, 15 and day 22 after start of treatment